CLINICAL TRIAL: NCT06870474
Title: Psychoeducational Intervention Against Support Groups for Caregivers: A Randomised Controlled Trial of Its Effectiveness
Brief Title: Psychoeducational Intervention Against Support Groups for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Sara Jiménez García-Tizón, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 454
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: dementia; effectiveness; family caregiver; psychoeducational intervention; support groups
MeSH Terms: conditions — Dementia | interventions — Self-Help Groups; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psychoeducational intervention (Experimental): The content was based on prior interventions, considering the caregivers' active involvement, adapting to their specific needs, addressing multiple areas of need, sporadic interventions over the course of the care, and the priority-based adjustment of the intensity or approach. This structure was adopted in all the sessions: 1) Review of homework, 2) Theoretical content, 3) Practical application of theoretical content, 4) Assignment of homework, and 5) Queries (see Table S1 of the supplementary material). The intervention involves eight 90-minute sessions held on a weekly basis
  Interventions: Behavioral: Psychoeducational intervention
- Support group (Placebo Comparator): In the sessions, caregivers share concerns and experiences with other group members, expressing feelings and fears. There is reciprocity, as they are listened to, but at the same time information is provided, ideas, strategies and skills are shared to face daily caregiving situations. The sessions are not structured, on the contrary, the topics are proposed and developed by the caregivers and the professional has only a moderating role. The intervention involves eight 90-minute sessions held on a weekly basis.
  Interventions: Behavioral: Support group
- Control group (Active Comparator): Caregivers were not subject to any intervention. They received the psychoeducational intervention once the study had ended.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Psychoeducational intervention — The psychoeducational intervention has the aim of improving quality of life, problem-solving and social skills, leisure time, self-efficacy and social support of caregivers; and decreasing their depressive symptomology, dysfunctional thoughts, burden and stress. Both mediator and outcome variables will be contemplated.
  Arms: Psychoeducational intervention
Behavioral: Support group — This intervention is a placebo group. It has the typical structure and characteristics of this type of intervention
  Arms: Support group
Behavioral: Control group — Participants were not subject to any intervention. They received the psychoeducational intervention once the study had ended.
  Arms: Control group

SUMMARY:
Background: To explore the effectiveness of a psychoeducational intervention against support groups and the usual care in caregivers. Providing care involves major changes in the lives of caregivers, with far-reaching repercussions. There is evidence that acting upon its mediator variables reduces its effects.

Methods: A randomised controlled trial will be carried out. The study will be conducted at the Faculty of Psychology of the University of Salamanca (USAL) in Spain. Family caregivers of people with dementia will participate in this study. The participants will be divided into three groups: the intervention group (IG), which will undergo a psychoeducational intervention programme, the support group (SG) (control group - placebo), which will undergo a support group intervention programme, and the control group-waiting lists (CG), which will only be assessed at the different measurements points, and after the end of the programme they will be offered the intervention of the experimental group. The programme (IG) will comprise eight sessions over a period of two months. All participants will be assessed at the outset and conclusion of the study, as well as after three and six months, during which time data regarding their socio-demographic characteristics and responses to the different scales will be collected. Both mediator and negative outcome variables will be assessed.

Discussion: Effective interventions need to be developed to improve the biopsychosocial state of caregivers. The presented psychoeducational intervention may help family caregivers because it could be more effective than others. The psychoeducational intervention has the aim of improving quality of life, problem-solving and social skills, leisure time, self-efficacy and social support of caregivers; and decreasing their depressive symptomology, dysfunctional thoughts, burden and stress.

ELIGIBILITY:
Inclusion Criteria:

* Be the main caregiver of a family member with dementia, either as a spouse or as an offspring.
* No previous involvement in studies/programmes like this one.
* The family member lives at home (not institutionalised).

Exclusion Criteria:

* Not be the main caregiver of a family member with dementia, either as a spouse or as an offspring.
* Previous involvement in studies/programmes like this one.
* The family member not lives at home (the family member is institutionalised).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Quality of life. The World Health Organization Quality of Life Assessment - AGE (WHOQOL-AGE) | Baseline; after 8 weeks; 3 and 6 months follow up
  It was assessed using the World Health Organization Quality of Life Assessment - AGE (WHOQOL-AGE). It contains 13 items in a Likert-type format with five options consisting of a combination of bipolar and unipolar responses. A higher score corresponds to a better quality of life
Stress. The Perceived Stress Scale (PSS) | Baseline; after 8 weeks; 3 and 6 months follow up
  Use was made of the Perceived Stress Scale (PSS). It consists of 14 items which assesses the level of stress the subject has perceived over the past month (from 0 = never to 4 = very often). The higher the direct score recorded, the higher the level of perceived stress.
Depressive symptomology. The Center for Epidemiologic Studies-Depression Scale (CES-D) | Baseline; after 8 weeks; 3 and 6 months follow up
  This was assessed through the Center for Epidemiologic Studies-Depression Scale (CES-D). It consists of 20 items which assess whether an individual has manifested any of the symptoms of depression during the preceding week (from 0 = rarely or never to 3 = mostly or all the time). A higher score corresponds to a greater depressive symptomology .
Burden. The Caregiver Burden Interview (CBI) | Baseline; after 8 weeks; 3 and 6 months follow up
  It was assessed using the Caregiver Burden Interview (CBI). It consists of 22 items which measures the extent to which caregivers perceive that their duties put a burden on their health, personal and social lives, finances, and emotional wellbeing (from 1 = never through to 5 = almost always). A higher score signals a greater burden.
Dysfunctional thoughts. Dysfunctional Thoughts Questionnaire. | Baseline; after 8 weeks; 3 and 6 months follow up
  The assessment used the Dysfunctional Thoughts Questionnaire. It measures the thoughts, opinions, values and attitudes of the caregivers of dependent elderly people (from 0 = completely disagree to 4 = completely agree) through 16 items. A higher score indicates the greater presence of obstacles for properly coping with caregiving.
Social support. The Psychosocial Support Questionnaire (PSQ) | Baseline; after 8 weeks; 3 and 6 months follow up
  This involved an adapted version of the Psychosocial Support Questionnaire (PSQ). It consists of six items (from 0 = never to 3 = always). The higher the score, the greater the perception of psychosocial support.
Social Skills. Social Skills Scale. | Baseline; after 8 weeks; 3 and 6 months follow up
  It was used the Social Skills Scale. It rates assertive behaviour and social skills (from 1 = it does not reflect me at all; it hardly ever happens to me, or I would not do it, to 4 = I completely agree and I would feel this way or act accordingly in most cases) through 33 items. The higher the global score, the greater the social skills.
Self-efficacy in caregiving. The Revised Scale for Caregiving Self-Efficacy (RSCSE). | Baseline; after 8 weeks; 3 and 6 months follow up
  The assessment used the Revised Scale for Caregiving Self-Efficacy (RSCSE). It assesses caregivers' own measure of their perceived self-efficacy for caregiving tasks through 15 items. It contains three subscales: Obtaining Respite, Responding to Disruptive Patient Behaviour, and Controlling Upsetting Thoughts. High scores reflect a significant level of self-efficacy.
Rewarding activities. The Leisure Time Satisfaction (LTS) scale | Baseline; after 8 weeks; 3 and 6 months follow up
  This was assessed thought an adapted version of the Leisure Time Satisfaction (LTS) scale. It consists of six items related to different leisure activities. It measures the frequency of performance (from 0 = not at all to 2 = a lot for) and the degree of satisfaction (from 0 = not at all satisfied to 2 = very) with it regarding rewarding activities in the past month. These are two scales with the same items. Higher scores correspond to a greater frequency and satisfaction with these activities.
Problem-solving skills. The Social Problem-Solving Inventory-Revised (SPSI-R-25) | Baseline; after 8 weeks; 3 and 6 months follow up
  This involved the Spanish version of the short form of the Social Problem-Solving Inventory-Revised (SPSI-R-25). It measures problem-solving skills (from 0 = not at all true to 4 = completely true). Higher scores indicate better social problem-solving.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, University of Salamanca, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No